CLINICAL TRIAL: NCT05400122
Title: A Phase Ib Study to Evaluate Safety and Persistence of ex Vivo Expanded Universal Donor NK Cells in Combination With IL-2 and TGFbeta Receptor I Inhibitor Vactosertib in Patients With Locally Advanced/Metastatic Colorectal Cancer, Gastric/Esophageal Cancer, and Relapsed/Refractory Hematologic Malignancies
Brief Title: Natural Killer (NK) Cells in Combination With Interleukin-2 (IL-2) and Transforming Growth Factor Beta (TGFbeta) Receptor I Inhibitor Vactosertib in Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs unavailable
Sponsor: David Wald (Other)
Responsible Party: Sponsor-Investigator, David Wald, IND Holder, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6Y21
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Hematologic Malignancy; Rectum Cancer; Acute Myeloid Leukemia; Myelodysplastic Syndromes; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Myeloproliferative Syndrome; Plasma Cell Myeloma; Gastric Cancer; Esophageal Cancer; Esophagus Cancer; Gastric Cancer, Metastatic; Unresectable Esophageal Cancer; Metastatic Esophageal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Hematologic Neoplasms; Rectal Neoplasms; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Stomach Neoplasms; Esophageal Neoplasms; Neoplasm Metastasis | interventions — vactosertib; fludarabine phosphate; Cyclophosphamide; Interleukin-2; aldesleukin; IL32 protein, human

STUDY DESIGN:
Intervention Model Description: Approximately 12 subjects will be enrolled in this trial and all will receive a preparative regimen consisting of lymphodepleting chemotherapy agents followed by two infusions of ex vivo-expanded NK cells in combination with vactosertib and IL-2 (Proleukin®).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Infusion (Experimental): Preparative Regimen Administration:
  * Fludarabine will be given at a dose of 30mg/m2 intravenously daily
  * Cyclophosphamide will be given at a dose of 500mg/m2 intravenously daily
  Investigational Agent Administration:
  * NK Cell Product will be given per institutional standard of care (at a rate no faster than 250mL per hour or 3-4 ml per minute) as two doses by intravenous infusion on Days 0 (+2 days acceptable) and 14 (+/- 3 days acceptable)
  * IL-2 will be administered at a flat dose of 2.2 million IU subcutaneously starting on the same day as the first NK cell infusion and will be administered three times weekly (dose level 1) or twice weekly (dose level -1) for up to four weeks total
  * Vactosertib will be administered at a dose of 200mg once daily for 5 consecutive days per week, for up to four weeks total.
  Interventions: Drug: Vactosertib; Drug: Fludarabine Phosphate; Drug: Cyclophosphamide; Drug: IL-2; Drug: Natural Killer Cells

INTERVENTIONS:
Drug: Vactosertib — Vactosertib is a highly selective, potent inhibitor of the protein serine/threonine kinase activity of transforming growth factor (TGF)-β receptor type 1 (TGFBR1; also known as activin receptor-like kinase 5 [ALK5]). Vactosertib inhibits the phosphorylation of the ALK5 substrates Smad2 and Smad3, as well as the intracellular signaling of TGF-β.
  Other Names: TEW-7197; EW-7197; EW7197
Drug: Fludarabine Phosphate — Fludarabine phosphate is rapidly dephosphorylated to 2-fluoro-ara-A and then phosphorylated intracellularly by deoxycytidine kinase to the active triphosphate, 2-fluoroara-ATP. This metabolite appears to act by inhibiting DNA polymerase alpha, ribonucleotide reductase and DNA primase, thus inhibiting DNA synthesis.
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide is an alkylating agent that prevents cell division by cross-linking DNA strands and decreasing DNA synthesis. It is a cell cycle phase nonspecific agent. Cyclophosphamide also possesses potent immunosuppressive activity.
  Other Names: Cytoxan; 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: IL-2 — Proleukin® (aldesleukin) has been shown to possess the biological activities of human native interleukin-2. In vitro studies performed on human cell lines demonstrate the immunoregulatory properties of Proleukin, including: a) enhancement of lymphocyte mitogenesis and stimulation of long-term growth of human interleukin-2 dependent cell lines; b) enhancement of lymphocyte cytotoxicity; c) induction of killer cell (lymphokine-activated (LAK) and natural (NK)) activity; and d) induction of interferon-gamma production.
  The in vivo administration of Proleukin in animals and humans produces multiple immunological effects in a dose dependent manner. These effects include activation of cellular immunity with profound lymphocytosis, eosinophilia, and thrombocytopenia, and the production of cytokines including tumor necrosis factor, IL-1 and gamma interferon. In vivo experiments in murine tumor models have shown inhibition of tumor growth
  Other Names: Proleukin
Drug: Natural Killer Cells — Adoptive NK cell therapy has demonstrated the potential for cancer immunotherapy in various malignancies with particular potential in hematologic malignancies including acute myeloid leukemia (AML), and colon cancer [14, 19-23]. This therapeutic approach is extremely well tolerated in patients even when massive numbers of cells are utilized (~109 NK cells/kg). In fact, studies suggest that high doses of NK cells are not only well tolerated but have potential to lead to higher levels of efficacy.

SUMMARY:
One of the ways that cancer grows and spreads is by avoiding the immune system.NK cells are immune cells that kill cancer cells, but are often malfunctioning in people with colorectal cancer and blood cancers. A safe way to give people with colorectal cancer and blood cancers fresh NK cells from a healthy donor has recently been discovered. The purpose of this study is to show that using two medicines (vactosertib and IL-2) with NK cells will be safe and will activate the donor NK cells. NK cells and vactosertib are experimental because they are not approved by the Food and Drug Administration (FDA). IL-2 (Proleukin®) has been approved by the FDA for treating other cancers, but the doses used in this study are lower than the approved doses and it is not approved to treat colorectal cancer or blood cancers.

DETAILED DESCRIPTION:
The goal of our study is to demonstrate that natural killer (NK) cells from non- HLA-matched donors can be safely infused into patients with colorectal cancer, patients with gastric or esophageal cancer, and patients with relapsed/refractory hematologic malignancies in combination with IL-2 and the oral TGFβ receptor I inhibitor vactosertib to improve the persistence of donor NK cells.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have one of the following:

  * Histologically confirmed locally advanced or metastatic colon or rectal adenocarcinoma
  * Histologically confirmed locally advanced or metastatic gastric, gastroesophageal junction, or esophageal adenocarcinoma
  * Relapsed or refractory hematologic malignancy
  * Acute myeloid leukemia with measurable residual disease (MRD) relapse
  * MRD relapse is defined as presence of ≥ 1 in 10-4 nucleated cells per European LeukemiaNet 2021 guidance [49]: (1) conversion of MRD negativity to MRD positivity, independent of the MRD technique, or (2) increase of MRD ≥1 log10 between any two positive samples measured in the same tissue (PB or BM) in patients with MRD-Low Level
  * Patients will be eligible if they have declined or are ineligible for standard treatment options and if there is no standard approach to curative therapy per NCCN guidelines. Patients with solid tumors must have had progression on at least one standard line of therapy.
  * Hematologic malignancies in the relapsed or refractory setting can include:

    * Acute myeloid leukemia
    * Myelodysplastic syndrome
    * Acute lymphoblastic leukemia
    * Chronic myeloid leukemia
    * Chronic lymphocytic leukemia
    * Non Hodgkin Lymphoma
    * Hodgkin Lymphoma
    * Myeloproliferative syndromes
    * Plasma cell myeloma
* Subjects must have recovered from acute toxicities of prior chemotherapy or stem cell transplant. Any prior non-hematologic vital organ toxicity (cardiac, pulmonary, hepatic, renal) of previous therapy must have resolved to grade 1 or less. Exceptions: Alopecia; subjects with chemotherapy-induced sensory neuropathy must have grade ≤ 3
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of NK cells in subjects ≤18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) Performance status ≤2
* Subjects must have normal organ and marrow function as defined below:

  * Serum total bilirubin <2 mg/dl. If known Gilbert syndrome, total bilirubin must be <3mg/dl
  * Aspartate aminotransferase (AST) < 2.5 X institutional upper limit of normal
  * Alanine Aminotransferase (ALT) < 2.5 X institutional upper limit of normal
  * Pulmonary function (DLCO) >40% of the expected value corrected for alveolar volume and hemoglobin
  * Serum Creatinine ≤ 1.5 X institutional upper limit of normal
  * Hemoglobin ≥ 7.5 g/dL
  * Absolute neutrophil count ≥ 1,250/mcL for colorectal cancer (CRC) patients or ≥ 1,000/mcL for patients with hematologic malignancies unless patient has bone marrow involvement of hematological malignancy
  * Platelet count ≥ 50,000/mcL; unless patient has bone marrow involvement of hematological malignancy
  * For patients with bone marrow involvement of hematologic malignancy, transfusion of blood products may be used to meet hemoglobin and platelet thresholds
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 4 weeks prior to study entry and for the duration of study participation. Women of child-bearing potential must have documented negative pregnancy test prior to start of lymphodepleting regimen. Child-bearing potential is defined by institutional standard.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.
* Subjects must have at least 3 weeks between last cytotoxic anti-neoplastic medication and initiation of preparative regimen.

Exclusion Criteria:

* Subjects receiving any other investigational agents
* Subjects requiring systemic corticosteroid therapy (10mg or less of prednisone or equivalent doses of other systemic steroids are permitted).
* Subjects for whom a potential 29-day delay in treatment will interfere with their potential therapeutic options
* Patients with active, untreated malignant involvement of the central nervous system (CNS) should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. If clinical suspicion for CNS involvement, head imaging will be necessary to document absence of active CNS involvement in patients with colorectal or esophagogastric cancer. Patients with hematologic malignancies who have undergone treatment for malignant involvement of the CNS must have no clinical evidence of residual CNS disease prior to study enrollment.
* History of allergic reactions to fludarabine or cyclophosphamide
* Subjects with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because cytotoxic agents used as part of the lymphodepleting regimen have the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with lymphodepleting chemotherapy, breastfeeding should be discontinued if the mother participates in the trial. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with chemotherapeutic agents. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy.
* Chronic active untreated hepatitis B or C infection. (Assessments should include Hepatitis B Surface Ab, Hepatitis B Surface Ag, Hepatitis B Core Ab - Total, Hepatitis B Core Ab, IGM, Hepatitis C Ab).
* Recipients of previous allogeneic transplants who have rash involving more than 10% body surface area attributed to graft versus host disease (GVHD). Stem cell transplant recipients will be excluded if they are still receiving immunosuppression including steroids for GVHD or have active GVHD in any organ (except for 10% BSA of skin, not requiring treatment).
* Subject who is taking prohibited medications when using vactosertib as following (refer to APPENDIX III). A minimal washout period of 5 half-lives for the following drugs is recommended prior to the first dosing.

  * Concurrent use of drugs or foods that are known strong CYP3A4 inhibitors including but not limited to grapefruit juice, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.
  * Concurrent use of drugs that are known potent CYP3A4 inducers including but not limited to phenytoin, rifampin, St. John's wort.
  * Concurrent use of drugs that are CYP3A4, CYP1A2, CYP2B6 substrates with narrow therapeutic indices including but not limited to theophylline, astemizole, cisapride, cyclosporine, dihydroergotamine, ergotamine, sirolimus, tacrolimus, terfenadine (astemizole, cisapride, and terfenadine have been withdrawn from the US market).
  * Concurrent use of drugs that are sensitive CYP3A4, CYP1A2, CYP2B6 substrates including but not limited to efavirenz, darunavir, dasatinib, everolimus, lopinavir, midazolam, sirolimus, ticagrelor.
* QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 12-lead ECGs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) | Within 28 days of NK cell infusion
  This will be defined as the incidence of Grade ≥ 2 treatment-related adverse events
Persistence of donor NK cells | 7 days post-treatment
  This will be defined as the presence of donor NK cells in recipient blood as determined by next-generation sequencing-chimerism at a frequency of >10%.

SECONDARY OUTCOMES:
Persistence of donor NK cells | 14 days post-treatment
  This will be defined as the presence of donor NK cells in recipient blood as determined by next-generation sequencing-chimerism at a frequency of >10%.
Persistence of donor NK cells | 21 days post-treatment
  This will be defined as the presence of donor NK cells in recipient blood as determined by next-generation sequencing-chimerism at a frequency of >10%.
Persistence of donor NK cells | 28 days post-treatment
  This will be defined as the presence of donor NK cells in recipient blood as determined by next-generation sequencing-chimerism at a frequency of >10%.
Clinical Response | 28 days post-treatment
  This will be defined as a change in size of measurable disease on CT scans (colorectal cancer) or by standard methods for hematologic malignancies (e.g. bone marrow biopsy for AML)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tomlinson, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States